CLINICAL TRIAL: NCT02209324
Title: Open-label Study of ASP2151 in Herpes Simplex Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M522101-J12
Record Dates: First submitted 2014-07-31; First posted 2014-08-05 (Estimated); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-02

CONDITIONS: Herpes Simplex
MeSH Terms: conditions — Herpes Simplex | interventions — ASP2151

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASP2151 (Experimental)
  Interventions: Drug: ASP2151

INTERVENTIONS:
Drug: ASP2151
  Other Names: 200 mg once daily

SUMMARY:
A multicenter, open-label study is conducted to evaluate the efficacy and safety of ASP2151 in patients with herpes simplex (recurrent labial/facial herpes and recurrent genital herpes and Kaposi varicelliform).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a rash associated with herpes simplex and a recurrent episode meeting the following criteria

   * Recurrent labial/facial herpes: Patients with at least 10 papulae or vesicles/pustules
   * Recurrent genital herpes: Patients with at least 5 papules or vesicles/pustules on the genital organs or in the genital and circumanal region
   * Kaposi varicelliform eruption: Patients with major skin symptoms of papulae or vesicles
2. Patients who can start receiving the study drug within 48 hours after onset of rash
3. Age: 16 years or older, but younger than 80 years

Exclusion Criteria:

1. Patients who are not expected to have an adequate response to oral antiviral medication.
2. Patients with two or more types of herpes simplex.
3. An extreme decline in immune function
4. Presence of serious complications
5. Patients found to meet any of the following conditions based on laboratory tests performed within 14 days before informed consent:

   * AST or ALT ≥ 2.5 x upper limit of normal
   * Platelet count < lower limit of normal
   * Serum creatinine ≥ 1.5 mg/dL
   * Creatinine clearance < 30 mL/min
6. Current or previous history of malignant tumor within 5 years before informed consent
7. Diagnosis of autoimmune disease

Ages: 16 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Sapporo Hokkaido Japan, Sapporo
  - Oota-ku Tokyo Japan, Tokyo
  - Yokohama Kanagawa Japan, Yokohama

RESULTS

PARTICIPANT FLOW:
Groups:
- ASP2151: 200mg once daily
Period: Overall Study
Arm/Group | ASP2151
Started | 275
Completed | 230
Not Completed | 45
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 14
Not completed — Withdrawal by Subject | 8
Not completed — Clinical laboratory value is ineligible on day 1 | 4
Not completed — Platelet count < LLN in Laboratory test | 7
Not completed — QT interval >-450 ms on measurement of an ECG | 5

BASELINE CHARACTERISTICS:
Population: Efficacy analysis set was defined as patients who were diagnosed with labial/facial herpes or recurrent genital herpes at the time of case registration, subsequently received the study drug at least once, and had any efficacy variable measured, except for those found not to have herpes simplex after study drug administration.
Arm/Group | ASP2151
Number analyzed (Participants) | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 247
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: year] | 39.2 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161
  Male | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 265
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 265
Region of Enrollment [Number; unit: participants]
  Japan | 265
Disease type [Count of Participants; unit: Participants]
  Recurrent labial / facial herpes | 191
  Recurrent genital herpes | 39
  Kaposi varicelliform eruption | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Healing by Day 8
Description: The percentage of participants achieving lesion healing by Day 8 of study treatment
Time Frame: 8 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | ASP2151
Number analyzed (Participants) | 265
Participants | 194

2. Secondary Outcome: Time to Healing
Description: The criteria for determining healing are as follows:
  1. A condition where all erythematous and papular lesions, vesicular and pustular lesions, and erosive and ulcerative lesions have been resolved, and either the complete resolution of crusts or the complete epithelialization beneath any remaining crusts has been achieved.
  2. In participants where no crust has formed, a condition characterized by the epithelialization of erosions/ulcers formation in mucosal lesions and potentially other affected areas.
  3. In participants where no vesicles or pustules have formed, a condition characterized by the complete resolution of all erythematous and papular lesions.
Time Frame: 29 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151
Number analyzed (Participants) | 265
day | 7 [5 to 8]

3. Secondary Outcome: Time to Complete Crusting
Description: The criteria for complete crust formation are outlined as follows:
  1. A condition where all erythematous and papular lesions, vesicular and pustular lesions, and erosive and ulcerative lesions have been resolved, and all rashes are crusted (epithelialization beneath is not required).
  2. In participants where no crust has formed, a condition characterized by the epithelialization of erosions/ulcers formation in mucosal lesions and potentially other affected areas.
  3. In participants where no vesicles or pustules have formed, a condition characterized by the complete resolution of all erythematous and papular lesions.
Time Frame: 29 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151
Number analyzed (Participants) | 265
day | 6 [5 to 8]

4. Secondary Outcome: Time to Virus Disappearance
Description: The day of viral disappearance is the first day on which the results of viral isolation continuously show 'HSV negative' until the final implementation day. The negative means that the results of the isolation and culture are negative, or the isolation and culture has not been performed due to complete crusting or healing of the lesion site.
Time Frame: 29 days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151
Number analyzed (Participants) | 265
day | 5 [3 to 6]

ADVERSE EVENTS:
Time Frame: 29 days
Description: The safety analysis population consisted of 271 participants, excluding four participants who were registered but never received the investigational drug.
Arm/Group | ASP2151
All-Cause Mortality (participants affected / at risk) | 0/271
Serious Adverse Events (participants affected / at risk) | 2/271
Other Adverse Events (participants affected / at risk) | 53/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ASP2151 (N=271)
Cellulitis of male external genitalorgan (Infections and infestations) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASP2151 (N=271)
Stomatitis (Gastrointestinal disorders) | 6
Nasopharyngitis (Infections and infestations) | 11
Folliculitis (Infections and infestations) | 6
Fibrin degradation products increased (Investigations) | 21
Alpha 1 microglobulin increased (Investigations) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes